CLINICAL TRIAL: NCT06466018
Title: Recherche de Biomarqueurs moléculaires et d'Imagerie Diagnostiques et Pronostiques Des Atteintes Oculaires associées à Des dérégulations Neurovasculaires : Cohorte Biocor
Brief Title: Research Into Diagnostic and Prognostic Molecular and Imaging Biomarkers of Ocular Disorders Associated With Neurovascular Deregulation: Biocor Cohort
Acronym: BIOCOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinact (Other)
Collaborators: Association CRO - Tous unis pour la vision (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-A02713-40
Record Dates: First submitted 2023-11-29; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Ocular Rosacea; Pachychoroid Disease
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ocular rosacea group (Experimental)
  Interventions: Diagnostic Test: Schirmer test paper
- Pachychoroid group (Experimental)
  Interventions: Diagnostic Test: Schirmer test paper
- Control group (Other)
  Interventions: Diagnostic Test: Schirmer test paper

INTERVENTIONS:
Diagnostic Test: Schirmer test paper — This paper is centrifuged and your tears are collected then frozen before analysis. We collect the fat from your tears by scraping the edge of your lower eyelid with small sterile tweezers. All surgical waste will be collected during eye surgeries only if you must have them.
  During each ocular surgical procedure, the vitreous, subretinal fluids and/or aqueous humor will eventually be recovered when required by the procedure. The rest of the blood samples, not used during diagnostic analyses, will be kept for later analyses.
  Tears will be collected using a non-invasive and painless method that takes around ten minutes. The tissues (connectiva, cornea, retina, epi-retinal membrane) which must have been removed when required by the surgical procedure will also be preserved.

SUMMARY:
BIOCOR is an interventional clinical trial whose main objectives are Objectif are identify molecular biomarker(s) of ocular rosacea and pachychoroid. Endpoints are : Correlation between pachychoroidosis (defined by choroidal phenotype parameters in OCT and autofluorescence) or the stage of ocular rosacea (ROSCO(29) definition) and biological markers selected on the basis of preclinical work (animal model) and by unbiased methods (proteomics, metabolomics, meibum lipidomics). The study of circulating, ocular and functional biomarkers would enable us to confirm our hypothesis and identify patients who could benefit from treatments that regulate the ANS and/or mineralocorticoid pathways.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 years of age, of European origin, with signed ± genetic consent
* Clear ocular media for OCT and autofluorescence imaging
* Signed consent form
* Be affiliated to a health insurance scheme
* Control patients are patients scheduled for cataract surgery or visual assessment.

Exclusion Criteria:

* High myopia > 6D
* Diabetic retinopathy, hereditary retinal dystrophy, untreated retinal detachment, choroidal ocular tumor, choroidal hemangioma
* Epithelial or stromal keratopathy other than ocular rosacea
* Corneal surgery less than 3 months old, keratoplasty
* Deprived of liberty or under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Clinical phenotype of ocular rosacea | Screening visit, visits A1, A2, and end-of-study visit
  * OSDI score
  * QoL score VF24 questionnaire
  * Stage and type of Rosacea
  * Blepharitis stage
  * Oxford score
  * Schirmer score
  * OSI Index
  * Meibomian meibography score
  * Quantification of corneal opacity and neovascularization by standardized score
  * Limbal insufficiency score
  * Clinical evolution under therapeutic effect
Pachychoroid clinical phenotype | From inclusion to end of study (Inclusion, year 1, year 2, year 3)
  * Measurement of total choroidal thickness
  * Measurement of choroidal vascular caliber
  * Measurement of foveolar avascular area
  * Calculation of fundus autofluorescence areas
  * Calculation of retinal non-perfusion areas
  * Cone counting

SECONDARY OUTCOMES:
Evolvolution of clinical profile of each phenotype in the cohort | From inclusion to end of study (Inclusion, year 1, year 2, year 3)
  Progression of limbic insufficiency (Deng grades) of ocular rosacea;
  * Ocular dryness (Oxford score, OSDI questionnaire);
  * Quantification of corneal nerves (density),
  * tear film (OSI score, Schirmer score, BUT score, OXFORD score),
  * meibomian glands (meibographic score);
  * variation in the thickness of the subfoveal choroid, a vascular index of the choroid quantified on analysis of the foveolar section in EDI;
  * Quantification of the surface area of epithelial atrophy on blue autofluorescence blue ;
Heart rate | At inclusion and end of study (Inclusion, year 3)
  * Measurement of static and dynamic heart rate variability (HRV) in patients and control group
  * Correlation of HRV with phenotypic stages and biological markers of interest

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of Ophthalmology, COCHIN Hospital, Paris, France